Strength training as a supplemental therapy for androgen deficiency of the aging male (ADAM): Study protocol for a three-arm clinical trial.

NCT03282682

23.03.2020

#### Aims

The overall aim of the trial is to examine the effect of a 12-week strength training program with and without TRT on body composition, physical function, selected biochemical markers of metabolic health, histological and molecular parameters and the quality of life of patients with ADAM.

## Study design

The study is a clinical trial with three arms comparing the effect of strength training with testosterone replacement therapy (ST + TRT), strength training alone (ST) on hypogonadal males and on a control group of healthy eugonadal males (HM), also engaged in strength training for 12 weeks.

## Trial status

At the time of the first submission of the protocol, the trial was in the phase of participant recruitment. The recruitment began in February 2017 and the last part of data collection is expected to end in August 2019.

### **Participants**

Subjects will be included from urological units at Department of Urology, University Hospital-Petrzalka, Bratislava, Slovakia; Department of Urology, Faculty of Medicine, Comenius University, Bratislava, Slovakia and 5. Department of Internal Medicine, Faculty of Medicine, Comenius University, Bratislava, Slovakia. The study will involve in total sixty-six male participants divided into three groups (n = 66): group 1, males with hypogonadism who are undergoing testosterone replacement therapy (TRT) (n=22); group 2, newly diagnosed males with hypogonadism without testosterone replacement therapy (NON-TRT) (n=22); group 3, healthy eugonadal men (HM) (n=22). The participants from all groups engaged in strength training. The volunteers are screened for testosterone levels before the start of the participation by the specialist.

The most important inclusion criteria for participation in the study from the patient population are age 40-60 years old, subjects with hypogonadism on TRT or newly diagnosed patients of hypogonadism. The hypogonadal patients fulfilling the criteria for study participation will be verified for low testosterone before entering the study. The same verification will take place at the end of the study. The most important exclusion criteria include regular strength training, conditions that are medical contraindications and prostate cancer or

abnormal serum PSA levels without adverse histological examination. All inclusion and exclusion criteria are listed in Additional file 1. In addition to written information, eligible subjects will be verbally informed about the study by their responsible urologist and the study officials before participation. TRT provided to patients is intramuscular (IM) injection of testosterone undecanoate (TU) at a dose of 1000 mg repeated every 12 weeks. Testosterone undecanoate (Nebido) is the only injectable form of testosterone used at the institutes of collaborating physicians of the study. According to our knowledge, this form of T at dose of 1000 mg is the most stable of all available preparations for 3 months' period, which is considered a standard treatment in Slovakia. Shorter-acting forms may cause more pronounced fluctuations in 24-hour circulating levels of testosterone. The participants will be asked to not change their habitual dietary intake and physical activity patterns. Participants will be asked to continue in physical activities as before, but any kind of regular physical activity, especially strength training or any other kind of weight training during the intervention will be also prohibited. The exclusion criteria reject any participant, who performed any kind of regular strength training one year prior to study.

# Strength training intervention

The strength training protocol will be a modified strength exercise program from Segal et al. [61] which was used in similar group of patients. The participants will perform 24 training sessions of strength training protocol with the frequency of two training sessions per week for 12 weeks. There will be at least 48 hours rest period between two subsequent training sessions (Monday and Thursday). The intervention will take place at the Faculty of Physical Education and Sport, Comenius University in Bratislava, Slovakia. All training sessions will be supervised and guided by professionals with university degree in sports training to ensure safety, correct technique and progression in training load, with a maximum of three participants per one trainer. The participants will be familiarised with the equipment and exercise technique one week before the start of the intervention. The technique corrections will be possible during the whole intervention if needed. Ten repetition maximum (RM) and 12RM diagnostic test for all exercises will be conducted during the first week of training intervention.

Each training session will include a 5-minute dynamic warm-up, consist of 10 exercises for approximately 30 seconds of each, and exercises will be focused on main muscle groups (Table 2).

Table 2: Dynamic warm-up

| Dynamic warm-up exercises | Number of repetitions |
|----------------------------|-----------------------|
| Walking low skip | 8 times each leg |
| Walking high knee skip | 8 times each leg |
| Walking knee to chest | 8 times each leg |
| Walking hamstring stretch | 6 times each leg |
| Walking lunge | 6 times each leg |
| Standing lateral lunge | 6 times each leg |
| Egyptian mobility exercise | 6 times each arm |
| External rotation exercise | 6 times each arm |
| Hip hinge exercise | 8 times |
| Air squat | 8 times |

The strength protocol exercises will be performed with free weights and on machines. The training program consist of six exercises for upper and lower body at an intensity of 60-80% (8 – 12RM: the load that induces technique failure in eight or twelve repetitions) of one-repetition maximum and takes approximately 60 minutes. The inability to perform full repetition will be assessed by a supervisor or by participants' feedback. The participants will be instructed to perform a concentric action for 2 seconds and immediately after an eccentric action also for 2 s. There will be 90 seconds rest period after each set. The same duration rest period will be between all of the exercises. The rest periods will be controlled by timer (The miniMAX, Gymboss, USA). The load will be added, if participant can complete prescribed number of repetition in each set of the exercise. More detailed strength training protocol can be seen in Table 3. During the first three weeks of the intervention, there will be one set in the beginning with light weight to focus on safety and technique. After that three more sets with weight close to 60 - 80% of 1RM will follow. After first three weeks, the number of sets will be increased to four.

Table 3: Strength training protocol

| Week | Number | of | Number | of | Number | of | Resistance | Rest | Tempo |
|---|---|---|---|---|---|---|---|---|---|
| | exercises | | sets | | repetitions | | | period | |

| 1 – 3. week | 3+3 (UB, LB) | 3 | 10-12 | 10-12RM | 90s | 2:0:2:1 |
|---------------|--------------|---|-------|---------|-----|---------|
| 4 – 6. week | 3+3 (UB, LB) | 4 | 10-12 | 10-12RM | 90s | 2:0:2:1 |
| 7– 9. week | 3+3 (UB, LB) | 4 | 6-8 | 6-8RM | 90s | 2:0:2:1 |
| 10 – 12. week | 3+3 (UB, LB) | 4 | 6-8 | 6-8RM | 90s | 2:0:2:1 |

UB – upper body, LB – lower body, RM – repetition maximum, Tempo – duration in seconds during the repetition - 2s (eccentric): 0s (end range of the motion): 2s (concentric): 1s (rest between repetitions in the starting position)

The exercises performed during every session will be: leg press, split squat, bench press. The exercises alternating through the week are knee extension with leg curl, seated row with seated pull down and incline dumbbell bench press (training equipment provided by KOHI Leopoldov, Slovakia and Technogym, Italia). Since unilateral exercises (e.g. one leg squats) develop similar magnitude of muscle activity with producing less load on the spine, thus they are safer [62], the split squats are chosen instead of regular squats. Prescribed exercises in the strength training protocol for every training sessions can be found in Table 4. Each session will be supervised by at least two professionals, who received strength training programme and record every repetition and set made in each session in an individual training plan. At the start of each session, the trainers will ask participants if they experienced any adverse events since the last session and record reported events. All adverse events during the training session will be written down into paper spread sheet and processed afterwards. Each training session will be monitored with an attendance list, with minimum 85% attendance during the study. Each session will be marked as successfully completed when at least 80% from the total volume and intensity of the training protocol planned for the particular training session is performed. If a participant will be unable to perform any of the exercises or sets, this will be recorded into a prepared training plan and the situation will be managed during the first week during familiarization with the training protocol. The appropriate alternative exercise will be considered depending on the restriction or participant's limitation.

Table 4: Training sessions, type of exercises and type of resistance

| 1st training session | Type of resistance | 2nd training session | Type of resistance |
|---|---|---|---|
| Split squat | Dumbbells | Bench press | Barbell |
| Bench press | Barbell | Split squat | Dumbbells |
| Leg press | Machine | Incline press | Dumbbells |
| Seated row | Machine | Leg press | Machine |
| Leg curl | Machine | Pull down | Machine |
| Lateral raise | Dumbbells | Knee extension | Machine |

#### Clinical outcomes

Clinical outcomes will be collected one week before the intervention (pre-intervention assessments) and one week after the intervention (post-training assessments). All outcomes, specific variables and assessments in each testing are listed in Additional file 2. All participants will be tested at the same time of the day, and asked to avoid caffeinated and alcohol beverages before the assessments

### Familiarization

To secure validity of the physical tests, all subjects undergo a session of familiarization 7 days prior to the intervention assessments. All sessions are performed based on the same guidelines, but after the familiarization session the load of each resistance exercise will be adjusted to match the expected maximum.

#### Primary outcome measure

Lean mass (LM)

The primary outcome of the study will be the change in lean mass (LM) measured by Dualenergy X-ray Absorptiometry (Hologic fan-beam bone densitometer Discovery QDR series). The changes in lower and upper body LM are analysed separately because of differences in androgen sensitivity in leg muscles compared to neck, chest and shoulder muscles [63]. Due to very similar results but greater participant comfort [63] we decided to use The National Health and Nutrition Examination Survey (NHANES) protocol, which required the participant to be positioned in a supine position in the middle of the densitometry table with head straight, space between the arms and torso, palms flat on the table, and feet together secured by a strap. The systematic review of Shiel et al. [64] showed a strong level of agreement as illustrated by high ICC's and CCC's between the Nana and NHANES positioning protocols, however systematic bias within limit of agreement plot and a large difference in 95% confidence limits indicates that the protocols should not be interchanged when assessing an individual.

#### Secondary outcome measures

Body composition

Other body composition parameters (fat mass, total body mass) will be measured at the same time so also the protocol is the same as with the primary outcome. The height will be measured by stadiometer and waist circumference will be measured by stretch-resistant tape that provides a constant 100 g tension. The body mass index is afterwards calculated and reported.

## Muscle strength

Muscle strength of lower extremities will be measured as force production during maximal voluntary contraction (MVC) isometric knee extension and isometric knee flexion knee dynamometer (ARS dynamometry, S2P ltd., Ljubljana, Slovenia). Each of the test will be performed 6 time with three practise trials and three recorded trials. For the first practise trial, participants will be instructed to achieve approximately 50% of the maximum, with 20 seconds rest period. The second and third practise trial will be performed at 80% of the maximum with 20 second rest periods. The last three trials will be performed with maximal voluntary effort and will be recorded. The best out of three will be taken for further analyses. Rest period during recorded trials will be 60 seconds. During the MVC, the participants will be asked to push/pull as strong as possible and hold for five seconds. Intra-session repeatability for MVC is the 5.7 CV % and 0,98 ICC. Additionally, with awareness of health issues (such as higher blood pressure) and because of a safety reasons, dynamic leg press 1RM (one repetition maximum) will be predicted from multiple repetition maximum testing [65].

For assessing the muscle strength of the upper extremities, the isometric MVC handgrip strength will be measured by Camry Digital Hand Dynamometer. The participant will stand upright and holds the dynamometer in the hand next to the body, with the minimal or none flexion in the elbow joint. The base of the handle will be on the first metacarpal, while the handle should rest on the middle of the four ringers. None of the body parts will be allowed to move. The test will be performed with three practise trials. First on 50% and the others on 80%

of their perceived maximum with 20 seconds' rest period. After that, three maximum trials with rest period of 60 seconds will be recorded and the best out of three will be taken for further analyses. The participants will be encouraged to give their maximum effort. The participant will squeeze the dynamometer for 5 seconds. After the test with dominant hand, the test will be performed for non-dominant hand.

### Cardio-respiratory fitness

Cardio-respiratory fitness will be measured by The Single Stage Treadmill Walking Test [66], where the participants will be asked to walk on Pro Treadmill (Woodway, USA). During the walking test, participants will wear same shoes they will use during the whole intervention. The speed during the test can be changed if needed. The procedure will be performed once and heartbeat will be tracked by heart rate monitor attached on the chest. VO<sub>2</sub>max will be calculated according the literature [66].

10-m preferred walk-speed and 10-m maximum walk-speed will be measured by timing gates WITTY GATE (MicroGate, Italy). Participants will walk 10 meters and the time will be measured for the intermediate 6 meters. This allow acceleration and deceleration. The gates will be placed on 2-meter mark and 8-meter mark. The timing starts when participant cross the first mark and stop when the 8-meter mark is crossed. There will be three trials for preferred and three trials for maximum walk-speed. The outcome measure will be velocity in meters per second calculated as mean of the three trials or the best trial from the preferred and maximum walk-speed test, respectively. Participants will be asked to perform at preferred walking speed first followedand then at the fastest walking speed possible.

### Psycho-social functioning

The general health status will be measured by The Short Form (36) Health Survey patient-reported survey of patient health (SF-36). In addition, clinically investigating the health-related quality of life (HRQoL) symptoms of aging men are measured by Aging Males' Symptom (AMS) Scale. The AMS scale had internal consistency [ $\alpha$  = 0.89 (95% CI 0.88-0.90)]; the mean alpha estimates across the AMS subscales ranged from 0.79 to 0.82. The AMS scale also had good test-retest reliability [r = 0.85 (95% CI 0.82-0.88]; the test-retest reliability coefficients of the AMS subscales ranged from 0.76 to 0.83 [67]. AMS is a standardized scale according to psychometric norms. Most of the currently available language versions were

translated following international standards for linguistic and cultural translation of quality of life scales. [68].

## Serological outcomes

Fasting morning venous blood will be taken after overnight (10-hour) fasting and 15 min rest from cubital vein from 8:00 am to 10:00 am [69] into closed system collection tubes containing beads coated with a clotting activator and polyacryl ester-gel (Sarstedt AG & Co, Germany). The blood will be centrifuged (3000g, 4°C, 10min) immediately after sampling to obtain EDTA plasma or they will be centrifuged (3000g, 4°C, 20min) after 30min at RT, to obtain serum. The haematological and biochemical parameters analyzed immediately will be haemoglobin, hematocrit, leucocytes, thrombocytes, glucose, urea, sodium, potassium, calcium, ALAT, total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride, testosterone, oestrogen, LH, FSH, SHBG, albumin, bilirubin, total protein, CRP, insulin and PSA. Plasma and serum aliquots (500 ul) will be stored at -20°C (analysis within 6 months) and at -80°C for the long term storage. Bioactive molecules (myokines, exerkines, released from skeletal muscle and/or other tissues) which could be associated with the adaptive response to exercise in all patients will be quantified.

### Muscle cellular outcomes

Muscle biopsies will be obtained from approximately 80% of the subjects included in the study. Subjects not willing to undergo biopsy are still eligible for trial participation.

With the subject in a supine position, a 5 mm Muscle Biopsy Cannula (Bergstrom-Stille, Sweden) with manual suction is used to obtain muscle samples (200 mg), under local anaesthesia (Lidocain 2%). Before the intervention, the biopsy will be obtained from the midsection of the right m. vastus lateralis, and after the intervention the biopsy will be obtained 3 cm proximal to the pre-intervention biopsy.

### Muscle fibre size and regulators of muscle fibre size

Muscle fiber size, measured as muscle fiber cross sectional area, represents the primary muscle cellular outcome. Secondary muscle cellular outcomes reflecting regulators of muscle fibre size

are a) number of myonuclei per muscle fiber b) number of satellite cells per muscle fiber, c) number of satellite cells and myonuclei positive for androgen receptors and d) proteins involved in muscle protein degradation (muscle breakdown). The number of satellite cells will be quantified on frozen muscle cross sections with a immunohistochemical protocol as described in Bjornsen et al. [70] (Pax7 + Laminin + DAPI).

Muscle fibre cross sectional area and regulators of muscle fibre size are analysed by immunohistochemistry on cross sections of muscle biopsies and by western blots and enzymelinked immunosorbent assay (ELISA) in muscle homogenate.

Muscle fibre cross sectional area is measured by cutting transverse serial sections of the muscle biopsy (8 µm thick) with a cryostat microtome (Microm, Germany) at -22°C and mounted on glass slides. Serial sections are immunohistochemically stained for fibre types (type I and type II) (used to measure muscle fibre cross sectional area), number of satellite cells, number of myonuclei and number of satellite cells and myonuclei positive for androgen receptors. Muscle fibre cross sectional area is measured for the different fibre types separately.

### Statistical Analysis

Normality of the data distribution will be assessed by comparing histogram of the sample data to a normal probability curve and outliers will be identified as values distant for more than  $3\sigma$  from the average. Normality will be further tested with Kolmogorov-Smirnov test if needed. Differences between normally distributed variables will be evaluated by the Analysis of variance with repeated measures and Bonferroni post-hoc test, differences between pre- and post-training values of the specific subpopulation will be evaluated with a paired Student's t-test. Non-normally distributed variables will be log transformed. Variables that could not be log transformed to normal distribution will be tested with non-parametric tests (Mann-Whitney test and Wilcoxon rank test).

Cohen's d will be used to calculate effect size (ES), represented by 'd' and interpreted as < 0.2 is a small, 0.2-0.8 is a moderate, and > 0.8 is a large effect size.

For studying the relationships between the various outcomes, the Pearson or Spearman correlation tests will be used.

All statistics were performed using a statistical software Statistical Package for the Social Sciences (SPSS) 21.0 (IBM Inc., Armonk, New York, U.S.,) and p values < 0.05 will be

considered significant. Data will be presented as means and standard deviations. Missing endpoint data will disqualify patient from the endpoint analysis. Missing single value, of training progression records will be replaced by the last observed value.

#### Background variables

Information about medical situation as time points for treatment and stage of symptoms are collected from the medical record. Past illnesses and other medical problems are also reported in the questionnaire.

#### Patients and public involvement

Patients (study participants) will be informed about the individual results of the baseline examination as well as on the primary and secondary outcomes of the study, in a form of individual consultation with a research team member.

Patients or public (patient organizations) were not involved in the development of the research question or study design. However, they will be asked to help with recruitment, and will also be involved in the conduct of the study with the power to shape (individualize) the training intervention according to individual preferences, prior experiences and medical conditions. Moreover, they will be involved in individualizing the follow-up intervention protocol, shaping thus the long-term exercise programme to increase its sustainability.

### Sample size

The pre-existing data from our previous 12-week exercise intervention study related to fat (5.6% decrease p=0.002) & lean body mass (1.8% increase, p=0.047, DXA) and that of maximal voluntary contraction force measured on linear leg-press (31% increase, p<0.0001, 1RM). Lean body mass was used to determine sample size for the population of the designed intervention study. The Type I error probability was set at 0.05 and the power to 0.90 and 0.95. Results indicate that 22 patients per group will be sufficient to detect exercise intervention related change of  $1,06 \pm 1,56$  kg (average  $\pm$  SD) of lean body mass at the power of 0.90, accounting for the 10% patients drop-out.

#### **Ethics and Dissemination**

This trial was approved by Ethics Committee of the University Hospital in Bratislava, Slovakia (ref. trial number: 127/2017). All the participants will be fully informed on the study protocol risks and benefits and will provide the written informed consent prior entering the study. Participation in the trial is fully voluntary. Inability to comply with the study protocol will not affect the healthcare. Data will be stored and handled anonymously using the coding system complying with the General Data Protection Regulation 2016/679. All unexpected, serious adverse events will be reported to the study sponsor as well as to the relevant health insurance company within 7 days. The findings of this trial will be published in peer review journals, scientific conferences with main audience of healthcare professionals, healthcare providers, but also patients and their families. Trial was registered at ClinicalTrials.gov: NCT03282682.

### **AUTHORS' CONTRIBUTIONS**

MK, JC, TR, MS participated in the study design and drafted the manuscript, GB participated in the development of the intervention protocol, TR, BU and JU designed protocol for biological sample collection and processing, and will participate in biological material sampling & analyses. MP, ZK, JP, BK and PB provide access to patients. MK, MS, JC, JU and MK performed data analysis. All authors contributed to and approved the present manuscript.

#### Full references:

- 1. Florini J. Effects of testosterone on qualitative pattern of protein synthesis in skeletal muscle. Biochemistry 1970 Feb 17;9(4): 909-12.
- 2. Vingren JL. Testosterone physiology in resistance exercise and training: The up-stream regulatory elements. Sports Medicine 2010;40(12): 1037–1053.
- 3. Dandona P, Rosenberg MT. A practical guide to male hypogonadism in the primary care setting. International Journal of Clinical Practice 2010;64(6): 682–696.
- 4. Kaufman JM, Vermeulen A. Declining gonadal function in elderly men. Bailliere's Clin Endocrinol Metab 1997;11(2): 289-309.
- 5. Tenover JS. Declining testicular function in aging men. Int J Impotence Res 2003; 15(Suppl 4): S3-8.

- 6. Feldman HA, Longcope C, Derby CA et al. Age trends in the level of serum testosterone and other hormones in middle-aged men: longitudinal results from the Massachusetts male aging study. J Clin Endocrinol Metab 2002; 87: 589–98.
- Wang C et al. Investigation, treatment and monitoring of late-onset hypogonadism in males: ISA, ISSAM, EAU, EAA and ASA recommendations. Eur J Endocrinol. 2008 Nov;159(5):507-14.
- 8. Bhasin S, Cunningham GR, Hayes FJ et al. Testosterone therapy in adult men with androgen deficiency syndromes: an endocrine society clinical practice guideline. J Clin Endocrinol Metab 2006; 91: 1995–2010.
- 9. Petak SM, Nankin HR, Spark RF et al. American Association of Clinical Endocrinologists Medical Guidelines for clinical practice for the evaluation and treatment of hypogonadism in adult male patients 2002 update. Endocr Pract 2002; 8:440–56.
- 10. Seftel A. Male hypogonadism. Part II: etiology, pathophysiology, and diagnosis. Int J Impot Res 2006; 18:223–8.
- 11. Carnegie Ch. 2004. Diagnosis of Hypogonadism: Clinical Assessments and Laboratory Tests. Rev Urol 2004;6(suppl 6): S3-S8.
- 12. Collier CP, Clark AF, Bain J et al. Functional testosterone: biochemical assessment of hypogonadism in men-report from a multidisciplinary workshop hosted by the Ontario Society of Clinical Chemists. The Aging Male: The Official Journal of the International Society for the Study of the Aging Male 2007; 10(4):211–216.
- 13. Arver S, Lehtihet M. Current guidelines for the diagnosis of testosterone deficiency. Horm Res 2009; 37: 5–20.
- 14. Morales A, Heaton JP, Carson CC III. Andropause: a misnomer for a true clinical entity. JUrol 2000; 163: 705–12
- 15. Tremblay RR, Gagne JM. Can we get away from serum total testosterone in the diagnosis of andropause? The Aging Male: The Official Journal of the International Society for the Study of the Aging Male 2005; 8(3–4): 147–150.
- 16. Shea JL et al. Free testosterone: clinical utility and important analytical aspects of measurement. Adv Clin Chem. 2014;63:59-84.
- 17. Smith MR, Finkelstein JS, McGovern FJ et al. Changes in body composition during androgen deprivation therapy for prostate cancer. J Clin Endocrinol Metab. 2002; 87:599–603.

- 18. Michael H, Härkönen PL, Väänänen HK, et al. Estrogen and Testosterone Use Different Cellular Pathways to Inhibit Osteoclastogenesis and Bone Resorption. Journal of Bone and Mineral Research 2005; 20:2224–2232.
- 19. Hak AE, Witteman JC, de Jong FH et al. Low levels of endogenous androgens increase the risk of atherosclerosis in elderly men: the Rotterdam study. J Clin Endocrinol Metab 2002; 87: 3632–9.
- 20. Allan CA, McLachlan RI. Age-related changes in testosterone and the role of replacement therapy in older men. Clinical Endocrinology 2004; 60(6): 653–670.
- 21. Fink JE, Hackney AC, Matsumoto M et al. Mobility and Biomechanical Functions in the Aging Male: Testosterone and the Locomotive Syndrome. Aging Male. 2018 Sep 29:1-8.
- 22. Mäkinen JI, Perheentupa A, Irjala K, et al. Endogenous testosterone and serum lipids in middle-aged men. Atherosclerosis 2008; 197:688–693.
- 23. Schwarz ER, Willix R. Impact of a physician-supervised exercise-nutrition program with testosterone substitution in partial androgen-deficient middle-aged obese men. Journal of Geriatric Cardiology 2011;8(4): 201–206.
- 24. Grossmann M, Thomas MC, Panagiotopoulos S et al. Low testosterone levels are common and associated with insulin resistance in men with diabetes. J Clin Endocrinol Metab 2008; 93:1834-40.
- 25. Ding EL, Song Y, Malik VS, Liu S. Sex differences of endogenous sex hormones and risk of type 2 diabetes: a systematic review and meta-analysis. JAMA 2006; 295:1288–1299
- 26. Rosario ER, Chang L, Stanczyk FZ et al. Age-Related Testosterone Depletion and the Development of Alzheimer Disease. JAMA 2004;292(12):1431-1432.
- 27. Moffat SD, Zonderman AB, Metter EJ et al. Longitudinal assessment of serum free testosterone concentration predicts memory performance and cognitive status in elderly men. J Clin Endocrinol Metab 2002; 87: 5001–5007.
- 28. Moffat SD1, Zonderman AB, Metter EJ et al. Free testosterone and risk for Alzheimer disease in older men. Neurology 2004;62(2):188-93.
- 29. Wang C, Swerdloff RS, Iranmanesh A et al. Testosterone Gel Study Group. Transdermal testosterone gel improves sexual function, mood, muscle strength and body composition parameters in hypogonadal men. J Clin Endocrinol Metab, 2000; 85:2839–53.
- 30. Page ST, Amory JK, Bowman FD, et al. Exogenous testosterone (T) alone or with fi nasteride increases physical performance, grip strength, and lean body mass in older men with low serum T. J Clin Endocrinol Metab, 2005; 90:1502–10.

- 31. Kapoor D, Aldred H, Clark S et al. Clinical and biochemical assessment of hypogonadism in men with type 2 diabetes: correlations with bioavailable testosterone and visceral adiposity. Diabetes Care 2007; 30:911–17.
- 32. Borst, SE, Mulligan T. Testosterone replacement therapy for older men. Clinical Interventions in Aging 200; 2(4), 561–566.
- 33. Nair KS, Rizza RA, O'Brien P et al. DHEA in elderly women and DHEA or testosterone in elderly men. N Engl J Med 2006, 355:1647–59.
- 34. Brill K, Weltman AL, Gentili A et al. Single and combined effects of growth hormone and testosterone administration on measures of body composition, physical performance, mood, sexual function, bone turnover, and muscle gene expression in healthy older men. J Clin Endocrinol Metab 2002 87:5649–57.
- 35. Clague JE, Wu FC, Horan MA. Difficulties in measuring the effect of testosterone replacement therapy on muscle function in older men. Int J Androl 1999; 22:261–5.
- 36. Kenny AM, Kleppinger A, Annis K et al. 2010. Effects of transdermal testosterone on bone and muscle in older men with low bioavailable testosterone levels, low bone mass, and physical frailty. J Am Geriatr Soc. 2010; 58(6):1134–1143.
- 37. Snyder PJ, Peachey H, Hannoush P et al. Effect of testosterone treatment on body composition and muscle strength in men over 65 years of age. J Clin Endocrinol Metab 1999; 84: 2647–2653.
- 38. Zitzmann M, Nieschlag E. Androgen receptor gene CAG repeat length and body mass index modulate the safety of long-term intramuscular testosterone undecanoate therapy in hypogonadal men. J Clin Endocrinol Metab 2007; 92: 3844–53.
- 39. Lasaite L, Ceponis J, Preiksa RT et al. Effects of two-year testosterone replacement therapy on cognition, emotions and quality of life in young and middle-aged hypogonadal men. Andrologia 2017; 49(3).
- 40. Hildreth, KL, Barry DW, Moreau KL et al. Effects of testosterone and progressive resistance exercise in healthy, highly functioning older men with low-normal testosterone levels. The Journal of Clinical Endocrinology and Metabolism 2013; 98(5), 1891–1900.
- 41. Permpongkosol S, Khupulsup K, Leelaphiwat S et al. Effects of 8-Year Treatment of Long-Acting Testosterone Undecanoate on Metabolic Parameters, Urinary Symptoms, Bone Mineral Density, and Sexual Function in Men With Late-Onset Hypogonadism. The Journal of Sexual Medicine 2016; 13(8), 1199–1211.
- 42. Bhasin S, Buckwalter JG. Testosterone supplementation in older men: a rational idea whose time has not yet come. J Androl. 2001 Sep-Oct;22(5):718-31.

- 43. Barrett-Connor E, Goodman-Gruen D, Patay B. Endogenous sex hormones and cognitive function in older men. J Clin Endocrinol Metab. 1999 Oct;84(10):3681-5.
- 44. Azad N, Pitale S, Barnes WE et al. Testosterone treatment enhances regional brain perfusion in hypogonadal men. J Clin Endocrinol Metab. 2003 Jul;88(7):3064-8.
- 45. Moffat SD, Zonderman AB, Metter EJ, et al. Longitudinal assessment of serum free testosterone concentration predicts memory performance and cognitive status in elderly men. J Clin Endocrinol Metab. 2002 Nov;87(11):5001-7.
- 46. McIntyre RS, Mancini D, Eisfeld BS et al. Calculated bioavailable testosterone levels and depression in middle-aged men. Psychoneuroendocrinology. 2006 Oct;31(9):1029-35. Epub 2006 Sep 5.
- 47. Kang DY, Li HJ. The effect of testosterone replacement therapy on prostate-specific antigen (PSA) levels in men being treated for hypogonadism: a systematic review and meta-analysis. Medicine (Baltimore). 2015 Jan;94(3): e410.
- 48. Loeb S, Folkvaljon Y, Damber JE et al. Testosterone Replacement Therapy and Risk of Favorable and Aggressive Prostate Cancer. J Clin Oncol. 2017 May 1;35(13):1430-1436.
- 49. Boyle P, Koechlin A, Bota M, et al. Endogenous and exogenous testosterone and the risk of prostate cancer and increased prostate-specific antigen (PSA) level: a meta-analysis. BJU Int. 2016 Nov;118(5):731-741.
- 50. Cui Y, Zong H, Yan H, et al. The effect of testosterone replacement therapy on prostate cancer: a systematic review and meta-analysis. Prostate Cancer Prostatic Dis. 2014 Jun;17(2):132-43.
- 51. Matsumoto AM. Andropause: clinical implications of the decline in serum testosterone levels with aging in men. J Gerontol A Biol Sci Med Sci 2002; 57:M76–99.
- 52. Bhasin S, Woodhouse L, Casaburi R et al. Older men are as responsive as young men to the anabolic effects of graded doses of testosterone on the skeletal muscle. Journal of Clinical Endocrinology and Metabolism 2005; 90(2), 678–688.
- 53. Rhoden EL, Morgentaler A. Risks of testosterone replacement therapy and recommendations for monitoring. N Engl J Med. 2004; 350:482-492.
- 54. Crewther B, Keogh J, Cronin J, Cook C. Possible stimuli for strength and power adaptation: acute hormonal responses. Sports Med 2006; 36:215–238.
- 55. Kraemer WJ, Marchitelli L, Scott GE et al. Hormonal and growth factor responses to heavy resistance exercise protocols. J Appl Physiol 1990; 69:1442–1450.

- 56. Newton RU, Taaffe DR, Spry N. et al. Can exercise ameliorate treatment toxicity during the initial phase of testosterone deprivation in prostate cancer patients? Is this more effective than delayed rehabilitation? BMC Cancer 2012;12:432.
- 57. Gardner JR, Livingston PM, Fraser SF. Effects of exercise on treatment-related adverse effects for patients with prostate cancer receiving androgen-deprivation therapy: A systematic review. Journal of Clinical Oncology 2014;32(4): 335–346.
- 58. Fink J, Schoenfeld BJ, Nakazato K. The role of hormones in muscle hypertrophy. Phys Sportsmed. 2018 Feb;46(1):129-134.
- 59. Glintborg D, Christensen LL, Kvorning T et al. Differential effects of strength training and testosterone treatment on soluble CD36 in aging men: Possible relation to changes in body composition. Scand J Clin Lab Invest. 2015;75(8):659-66.
- 60. Cho DY, Yeo JK, Cho SI et al. Exercise improves the effects of testosterone replacement therapy and the durability of response after cessation of treatment: a pilot randomized controlled trial. Asian J Androl. 2017;19(5):602-607.
- 61. Segal RJ, Reid RD, Courneya KS et al. Resistance exercise in men receiving androgen deprivation therapy for prostate cancer. J Clin Oncol 2003; 21:1653-1659.
- 62. Eliassen W, Saeterbakken AH, van den Tillaar R. Comparison of bilateral and unilateral squat exercises on barbell kinematics and muscle activation. Int J Sports Phys Ther. 2018 Aug;13(5):871-881.
- 63. Kadi F. Adaptation of human skeletal muscle to training and anabolic steroids. Acta Physiol Scand Suppl 2000; 646:1-52.
- 64. Shiel F, Persson C, Furness J, et al. Dual energy X-ray absorptiometry positioning protocols in assessing body composition: A systematic review of the literature. J Sci Med Sport. 2018 Oct;21(10):1038-1044.
- 65. Reynolds JM, Gordon TJ, Robergs RA. Prediction of one repetition maximum strength from multiple repetition maximum testing and anthropometry. Strength Cond Res 2006;20(3):584-92.
- 66. Ebbeling CB, Ward A, Puleo EM et al. Development of a single-stage submaximal treadmill walking test. Med Sci Sports Exerc 1991;23(8):966-73.
- 67. Lee CP, Chiu YW, Chu CL, et al. A reliability generalization meta-analysis of coefficient alpha and test-retest coefficient for the aging males' symptoms (AMS) scale. Aging Male. 2016 Dec;19(4):244-253.

- 68. Heinemann LA, Saad F, Zimmermann T et al. The Aging Males' Symptoms (AMS) scale: update and compilation of international versions. Health Qual Life Outcomes. 2003 May 1;1:15.
- 69. Gonzalez-Sales M, Barriere O, Tremblay PO et al. Modelling Testosterone Circadian Rhythm in Hypogonadal Males: Effect of Age and Circannual Variations. The AAPS Journal 2016; 18(1), 217–227.
- 70. Bjørnsen T, Wernbom M, Kirketeig A et al. Type 1 Muscle Fiber Hypertrophy after Blood Flow-restricted Training in Powerlifters. Med Sci Sports Exerc. 2019 Feb;51(2):288-298.

## Funding statement

The study is funded by the Scientific Grant Agency of the Ministry of Education, Science, Research and Sport of the Slovak Republic and of the Slovak Academy of Sciences (VEGA) no. 1/0714/16.

# Competing interests statement

We declare that we have no significant competing financial, professional, or personal interests that might have influenced the performance or presentation of the work described in this manuscript.